CLINICAL TRIAL: NCT02325414
Title: Prevention of Bone Loss After Acute SCI by Zoledronic Acid: Durability, Effect on Bone Strength, and Use of Biomarkers to Guide Therapy
Brief Title: Prevention of Bone Loss After Acute SCI by Zoledronic Acid
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Thomas J. Schnitzer, Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: STU00098239; CDMRP-130125 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2014-12-21; First posted 2014-12-25 (Estimated); Results first posted 2021-06-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Spinal Cord Injury; Acute Spinal Cord Injury; Bone Loss; Osteoporosis
Keywords: Osteoporosis; Spinal Cord Injury; Bone Diseases; Metabolic Bone Diseases; Musculoskeletal Diseases; Spinal Cord Diseases; Central Nervous System Diseases; Nervous System Diseases; Nervous System; Wounds and Injuries; Bone Density Conservation Agents; Physiological Effects of Drugs; Pharmacologic Actions; Department of Defense
MeSH Terms: conditions — Spinal Cord Injuries; Bone Diseases, Metabolic; Osteoporosis; Bone Diseases; Musculoskeletal Diseases; Spinal Cord Diseases; Central Nervous System Diseases; Nervous System Diseases; Neurologic Manifestations; Wounds and Injuries | interventions — Zoledronic Acid; Diphosphonates; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Zol (Experimental): Intravenous infusion of zoledronic acid (zol) 5 mg at baseline.
  Interventions: Drug: Zoledronic acid
- Placebo (Experimental): Intravenous infusion of placebo at baseline.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zoledronic acid — Intravenous infusion of zoledronic acid 5 mg.
  Other Names: Reclast; Zometa; Bisphosphonate
  Arms: Zol
Drug: Placebo — Placebo (saline) infusion to match zoledronic acid
  Other Names: Saline
  Arms: Placebo

SUMMARY:
The overall objective of this study is to define an effective therapeutic approach, using currently available medication, to prevent or mitigate the loss of bone mass and bone strength that occurs after acute spinal cord injury.

DETAILED DESCRIPTION:
This is a randomized, double-blind placebo-controlled study of zoledronic acid to evaluate its efficacy and safety over a 2 year period for the prevention of bone loss and maintenance of bone strength in individuals with recent onset SCI (see diagram below). Subjects will be randomized at the baseline visit to receive either zoledronic acid or placebo. At the end of the first year of the study, each treatment group will be re-randomized to either zoledronic acid or placebo to evaluate the durability of response to zoledronic acid and the utility of serum bone markers to guide therapeutic decision making. DXA imaging, CT imaging and bone markers will be obtained at baseline, 3 months, 6 months, 12 months, 18 months and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* In-patient at Rehabilitation Institute of Chicago (RIC) or an outpatient who was recently discharged from RIC
* Males and females
* Age >/=18 years
* Medically stable in the opinion of subject's physiatrist
* SCI at within 120 days inclusive at time of screening
* SCI with inability to ambulate independently
* ASIA Impairment Scale (AIS) A, B, or C, at time of study entry
* Capable of positioning to have DXA performed
* Able to tolerate acetaminophen
* No known endocrinopathies (diabetes type 1 or 2 can be included)
* Normal TSH levels
* Normal 25-OH vitamin D levels (>/= 20 ng/ml) at baseline (subjects may be repleted)
* Normal calcium levels
* Normal renal function (creatinine <2.0 mg/dl)
* Well hydrated with adequate intake of liquids
* Able to return for all follow-up visits
* Capable of reading and understanding informed consent document
* Males and females of childbearing potential must be willing and able to use double barrier method of contraception for 2 months after having received study drug

Exclusion Criteria:

* Have Paget's disease of the bone
* Malignancy as a cause of acute SCI
* Have unexplained high levels of alkaline phosphatase in blood
* Any active gastrointestinal condition that results in malabsorption
* Poor dental hygiene or requirement for invasive dental procedure within two months prior to enrollment
* History of bone metastasis and skeletal malignancies
* History of alcoholism or drug abuse within the 2 years prior to study screening
* Other medical conditions that in the opinion of the investigator would preclude the subject from completing the study
* Elevated liver function tests >2x normal
* Currently being prescribed anti-convulsants at a dose or frequency that is determined to interfere with bone metabolism as determined by the investigator
* Currently being prescribed glucocorticoids, other than inhaled glucocorticoids
* Current or recent use any bone-active agents, including any bisphosphonate, raloxifene, hormone therapy (estrogen and estrogen/progestin), calcitonin or strontium-containing compounds within 60 days of screening.
* Pregnant, planning to become pregnant, or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2020-08-25 (Actual); Study Completion 2020-08-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J Schnitzer, MD, PhD, Principal Investigator — Northwestern University Feinberg School of Medicine
Locations (2):
- United States (2):
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Rehabilitation Institute of Chicago, Chicago, Illinois

REFERENCES:
- [Derived] Edwards WB, Haider IT, Simonian N, Barroso J, Schnitzer TJ. Durability and delayed treatment effects of zoledronic acid on bone loss after spinal cord injury: a randomized, controlled trial. J Bone Miner Res. 2021 Nov;36(11):2127-2138. doi: 10.1002/jbmr.4416. Epub 2021 Jul 29. PMID 34278611
- [Derived] Haider IT, Lobos SM, Simonian N, Schnitzer TJ, Edwards WB. Bone fragility after spinal cord injury: reductions in stiffness and bone mineral at the distal femur and proximal tibia as a function of time. Osteoporos Int. 2018 Dec;29(12):2703-2715. doi: 10.1007/s00198-018-4733-0. Epub 2018 Oct 17. PMID 30334093

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with acute SCI were recruited from the Shirley Ryan AbilityLab, formerly known as the Rehabilitation Institute of Chicago. Recruitment took place between February 2015 and February 2018.
Pre-assignment Details: After meeting eligibility, participants were randomized in a blinded fashion and received study drug at the baseline visit.
Groups:
- Zoledronic Acid: Intravenous infusion of zoledronic acid (zol) 5 mg at baseline.
- Placebo: Intravenous infusion of placebo (saline) at baseline.
Period: Overall Study
Arm/Group | Zoledronic Acid | Placebo
Started | 30 | 30
Completed | 22 | 24
Not Completed | 8 | 6
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Lost to Follow-up | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zoledronic Acid | Placebo | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 28 | 57
  >=65 years | 1 | 2 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.3 (15.9) | 38.2 (15.2) | 37.8 (15.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 3 | 12
  Male | 21 | 27 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 7 | 11
  Not Hispanic or Latino | 26 | 23 | 49
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 6 | 14
  White | 20 | 21 | 41
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60
Time Since Injury (Days) [Mean (Standard Deviation); unit: days] | 68.7 (28.5) | 62.7 (23.2) | 65.7 (25.9)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Bone Mass Density (BMD) in the Hip
Description: Percent change of bone mass density (BMD) in the total hip (as measured by DXA)
Time Frame: 0-12 months
Measure: Median (Inter-Quartile Range); unit: percent change in bone mass density
Arm/Group | Zoledronic Acid | Placebo
Number analyzed (Participants) | 30 | 30
percent change in bone mass density | -2.21 [-8.93 to 4.51] | -12.82 [-29.04 to 3.40]
Statistical Analysis 1: Comparison: Zoledronic Acid vs Placebo; Test type: Superiority; p = 0.05, Mixed Models Analysis; Median Difference (Final Values) = 10.61; One-year data analysis were carried out using linear mixed-effects models. Covariate adjustments for baseline value of the corresponding outcome and ambulatory status (measured by WISCI) were performed by fitting these variables as fixed factors. The repeated measures were addressed using participant identification as random intercepts in the model

2. Primary Outcome: Percent Change of Bone Mass Density (BMD) in the Femoral Neck
Description: Percent change of bone mass density (BMD) in the femoral neck (as measured by DXA)
Time Frame: 0-12 months
Measure: Median (Inter-Quartile Range); unit: percent change in bone mass density
Groups:
- Zoledronic Acid (Zol): Intravenous infusion of the study drug zoledronic acid (Zol) 5 mg at baseline.
- Placebo (Pla): Intravenous infusion of placebo at baseline.
  Placebo (Pla): saline
Arm/Group | Zoledronic Acid (Zol) | Placebo (Pla)
Number analyzed (Participants) | 30 | 30
percent change in bone mass density | -1.72 [-7.05 to 3.59] | -11.34 [-22.29 to -0.39]

3. Secondary Outcome: Percent Change in the Epiphyseal Integral Bone Mass Content (iBMC) of the Femur
Description: Percent change in the epiphyseal integral bone mass content (iBMC) of the femur, as collected by CT.
Time Frame: 0-12 months
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Zoledronic Acid (Zol) | Placebo (Pla)
Number analyzed (Participants) | 30 | 30
percent change | -9.6 [-31.02 to 11.82] | -22.90 [-50.72 to 4.92]

4. Secondary Outcome: Percent Change in the Metaphyseal Integral Bone Mass Content (iBMC) of the Femur
Description: Percent change in the metaphyseal integral bone mass content (iBMC) of the femur, as collected by CT
Time Frame: 0-12 months
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Zoledronic Acid (Zol) | Placebo (Pla)
Number analyzed (Participants) | 30 | 30
percent change | -4.73 [-13.83 to 4.37] | -8.88 [-19.12 to 1.36]

ADVERSE EVENTS:
Time Frame: Baseline - 12 month visit
Description: Adverse event collection began at the baseline visit, as soon as the participant received the first year study drug infusion. At each study visit, participants were asked about any changes to their health.
Groups:
- Zoledronic Acid: Intravenous infusion of the study drug zoledronic acid (Zol) 5 mg at baseline.
- Placebo: Intravenous infusion of placebo at baseline.
  Placebo (Pla): saline
Arm/Group | Zoledronic Acid | Placebo
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 8/30 | 9/30
Other Adverse Events (participants affected / at risk) | 28/30 | 22/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zoledronic Acid (N=30) | Placebo (N=30)
Acute Phase Response (General disorders) | 2 (2) | 0 (0) — Defined as a flu-like reaction beginning within 3 days after the study drug (Zol) infusion, and included some or all of the following symptoms: fever, chills, headaches, nausea, vomiting, loss of appetite, and/or bone, joint, or muscle pain.
Altered Mental Status (Psychiatric disorders) | 1 (2) | 0 (0)
Autonomic Dysreflexia (Nervous system disorders) | 0 (0) | 2 (2)
C. difficile Infection (Infections and infestations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Thrombus (Vascular disorders) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Exophoria with Intermittent Exotropia (Eye disorders) | 1 (1) | 0 (0)
Gas (Incidental finding on X-ray) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Immune Thrombocytopenic Purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neuropathy, new or worsened (Nervous system disorders) | 0 (0) | 1 (1)
Osteomyelitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle pain (Back) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Panic Attack (Psychiatric disorders) | 1 (1) | 0 (0)
Pressure Ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pyelonephritis (Renal and urinary disorders) | 0 (0) | 1 (1)
Septic Shock (Infections and infestations) | 1 (1) | 1 (1)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Traumatic Catheterization (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Urinary Tract Infection (Renal and urinary disorders) | 3 (4) | 5 (5)
Worsened Psychiatric Symptoms (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zoledronic Acid (N=30) | Placebo (N=30)
Acute Phase Response (General disorders) | 20 (20) | 3 (3) — Defined as a flu-like reaction beginning within 3 days after the study drug (Zol) infusion, and included some or all of the following symptoms: fever, chills, headaches, nausea, vomiting, loss of appetite, and/or bone, joint, or muscle pain.
Autonomic Dysreflexia (Nervous system disorders) | 3 (4) | 1 (1)
Burn (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Chills (General disorders) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Cough (General disorders) | 3 (3) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Fatigue/Weakness (General disorders) | 1 (1) | 2 (2)
Fever (General disorders) | 2 (2) | 3 (3)
Flu (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Fungal Infection (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Headache (General disorders) | 0 (0) | 2 (2)
Heterotopic Ossification, new or worsened (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Hypertension (Vascular disorders) | 3 (3) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Joint Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Neuropathy, new or worsened (Nervous system disorders) | 0 (0) | 2 (3)
Pressure Ulcer (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (4)
Spasticity, new or worsened (Nervous system disorders) | 2 (2) | 2 (2)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 8 (8)
Urinary Tract Infection (Renal and urinary disorders) | 15 (26) | 10 (19)
Worsened Depression Symptoms (Psychiatric disorders) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
The number of participants in the trial was limited, particularly during the second year in each subgroup. Additionally, the number of women studied was limited but was representative of the general sex distribution observed in people with spinal cord injury.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-06-28): https://cdn.clinicaltrials.gov/large-docs/14/NCT02325414/Prot_001.pdf
  • Statistical Analysis Plan (2020-06-17): https://cdn.clinicaltrials.gov/large-docs/14/NCT02325414/SAP_002.pdf